CLINICAL TRIAL: NCT03375996
Title: Evaluation of a Preoperative Pharmacological Protocol for Mydriasis in Femtosecond Laser-assisted Cataract Surgery
Brief Title: Evaluation of a Protocol of Pupil Dilation Before Laser-assisted Cataract Surgery
Acronym: MYFLACS
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO17111*
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cataract Surgery
MeSH Terms: interventions — Cyclopentolate; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FLACS group: Patient presenting cataract and scheduled for laser-assisted cataract surgery
  Interventions: Drug: cyclopentolate 0.5% eye drops

INTERVENTIONS:
Drug: cyclopentolate 0.5% eye drops — cyclopentolate 0.5% eye drops and measurement of the pupillary mydriasis (dilatation)

SUMMARY:
Laser-assisted cataract surgery is an innovative and growing procedure to improve the safety and results of modern cataract surgery. However, this technique faces to some obstacles: economics in the one hand due to the cost and time spent for the laser procedure before the conventional surgery, and technical in the other hand, especially due to some loss of pupil dilation during the surgery, which is highly important to ensure a perfect procedure. The present study aims at assessing a pharmacological protocol to maintain an accurate pupil dilation all along the surgery in order to improve the whole procedure.

DETAILED DESCRIPTION:
Femtosecond laser-assisted cataract surgery (FLACS) is a major surgical development that would allow systematization of surgery and even improved safety of the procedure. The development of this new surgical technique must now face certain obstacles, in particular (i) financial considering the extra cost generated by the use of the laser and (ii) technique due to the need to re-learn certain gestures and certain variations related to the laser procedure and more specifically the instability of the pupillary mydriasis (dilatation) during the actual surgery. The use of a systematic preoperative pharmacological mydriasis protocol should allow maximum intraoperative mydriasis to be maintained, allowing satisfactory surgery throughout the procedure. Several drugs or medical devices are now indicated in cataract surgery, but their effectiveness has not been specifically evaluated for the laser technique. This study could thus make it possible to validate or not a protocol of mydriasis that could make consensus in the future for the practice of FLACS.

ELIGIBILITY:
inclusion criteria :

* Patient with unilateral or bilateral cataract requiring a cataract surgery
* Patient scheduled for laser-assisted cataract surgery

exclusion criteria :

* Limitation due to laser procedure (little orbits, corneal scares, lack of pharmacological mydriasis at the inclusion visit)
* Subject with general medication influencing iris state and/or pupil dilation (alpha-agonist, psychotropic drugs)
* Subject unable to give informed consent
* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cataract scheduled for laser-assisted cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Pupil diameter > 6 mm all along the surgical procedure | Day 0
  a posteriori pupil measurement using the peroperative movie recorded via the operative microscope during each surgery.

SECONDARY OUTCOMES:
Pupil diameter variation at each time of the surgery | Day 0
Surgeon satisfaction | Day 0
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France